CLINICAL TRIAL: NCT05791929
Title: Image Features of LSCI and Thermography for Prediction of Healing Trajectory in Diabetic Foot Patients Affected by the First (or Successive) Ulcer: (MY-FOOT-B)
Brief Title: LSCI and Thermography in Diabetic Foot Patients Affected by Ulcer(s): (MY-FOOT-B)
Acronym: MY-FOOT-B
Status: Withdrawn | Type: Observational
Why Stopped: MY FOOT study proposal was submitted for the HORIZON-HLTH-2023-TOOL-05-03 call, but the project was not approved
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor
Other Study IDs: MY-FOOT-B
Record Dates: First submitted 2023-03-17; First posted 2023-03-30 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1; Ulcer Foot
Keywords: Diabetes; Ulcer foot; LSCI; Thermography
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1; Foot Ulcer; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this observational study is to predict healing at 26 weeks after the first visit in patients affected by the first ulcer, by means of combined data monitoring of Laser Speckle Contrast Imaging (LSCI) and temperature measurements during patient visits in hospital.

In order to achieve this objective, study aims to produce a logistic regression model and then evaluate its prognostic ability by means of the area under the curve (AUC) of the receiver-operating-characteristics (ROC) curve.

Patients with diabetes mellitus and suffering from ulcer and receiving health care will undergo regular microcirculatory measurements including LSCI scans in and around the ulcer location and thermography.

DETAILED DESCRIPTION:
The study aims to predict healing at 26 weeks after the first visit in patients affected by the first ulcer, by means of combined data monitoring of Laser Speckle Contrast Imaging (LSCI) and temperature measurements during patient visits in hospital.

In order to achieve this objective, the study aims to produce a logistic regression model and then evaluate its prognostic ability by means of the area under the curve (AUC) of the receiver-operating-characteristics (ROC) curve.

The variables evaluated for the model will include demographic and baseline characteristics of the patients, location and seriousness of the ulcer, alongside LSCI and temperature measurements at baseline and different timepoints. The development of the model will include a rigorous variables selection in order to produce a parsimonious model.

In the method proposed by Mennes, LSCI measurements at baseline, biological zero, post occlusion peak, and other parameters like non-invasive blood pressure measurements were individually evaluated as possible prognostic factors of healing trajectory at 26 weeks. All these parameters, when assessed at their highest possible value of sensibility and specificity, produced AUCs always inferior to 0.65. The highest value of AUC (0.625) was reached by toe pressure parameter when calculated using a threshold value of 54 mmHg.

From diagnostic literature, an AUC of ≥ 0.8 is considered excellent result, while an AUC < 0.7 is considered less than acceptable. Since the Mennes's method showed these results, study investigators set the AUC resulting from the model under the null hypothesis (H0) to be equal to 0.65. By including all these parameters, alongside the other mentioned variables, in a single prognostic model, study investigators expect to increase this prognostic ability. Therefore, in this study, investigators would like to detect an AUC ≥ 0.8 (H1). With these hypotheses, a power of 80%, a one-sided I type error of 5% and a prevalence of 43% of healed patients at 26 weeks, a total of 82 patients should be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* a confirmed diagnosis of type 1 or type 2 diabetes mellitus (more than 5 years from diagnosis),
* aged between 18 and 80 years,
* patients affected by one foot ulcer (defined as break of the skin of the foot that involves at least the epidermis and part of the dermis )
* signed informed consent.

Exclusion Criteria:

* having multiple foot ulcers,
* having an amputation of the forefoot or an amputation at a more proximal location of the foot (e.g., midfoot or hindfoot),
* severe foot infection (IWGDF grade 4),
* being incapacitated or undergoing cancer treatment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diabetes mellitus and suffering from ulcer and receiving health care at study participating hospitals
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-04-13 (Actual); Primary Completion 2023-10-10 (Estimated); Study Completion 2023-12-04 (Actual)

PRIMARY OUTCOMES:
Area Under ROC curve generated by the statistical model able to discriminate between healing and not healing ulcers | at 26 weeks after the first visit in patients affected by the first ulcer
  to discriminate between healing and not healing ulcers by means of combined data monitoring of Laser Speckle Contrast Imaging (LSCI) and temperature measurements during patient visits in hospital

SECONDARY OUTCOMES:
The predictive positive and negative value related to the score test, based of calculation of likelihood ratio. | at 26 weeks after the first visit in patients affected by the first ulcer
  The predictive positive and negative value related to the score test, based of calculation of likelihood ratio.
The AUC of the models estimated according to different sites of ulcers. | at 26 weeks after the first visit in patients affected by the first ulcer
  The AUC of the models estimated according to different sites of ulcers.

CONTACTS AND LOCATIONS:
Overall Officials: Cesare Miranda, MD, Principal Investigator — Pordenone Hospital

IPD SHARING:
Plan to Share IPD: No
There is a plan to make individual participant data (IPD) available to other researchers